CLINICAL TRIAL: NCT00278772
Title: "A Randomized, Double-Blind, Placebo-Controlled Study of Divalproex Extended Release Monotherapy in Ambulatory Bipolar Spectrum Disorder With Moderate-to- Severe Hypomania or Mild Mania"
Brief Title: Study of Divalproex Extended Release Monotherapy in Ambulatory Bipolar Spectrum Disorder With Moderate-to-Severe Hypomania or Mild Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Abbott (Industry); University of Cincinnati (Other)
Responsible Party: Susan McElroy, MD / Professor, Lindner Center of HOPE
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Miefert
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Bipolar Spectrum Disorder With Moderate-to- Severe Hypomania or Mild Mania
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): Divalproex
  Interventions: Drug: Divalproex
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Divalproex — oral, 15mg/kg/day - 30mg/kg/day
  Arms: 1
Other: Placebo — oral dose, placebo
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability, and efficacy of divalproex extended release compared to placebo (sugar pill without medication) in the treatment of bipolar disorder with moderate to severe hypomania or mild mania. Divalproex extended release is approved by the United States Food and Drug Administration (FDA) for the treatment of epilepsy and for prevention of migraine headaches.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of divalproex extended release (DPX-ER) monotherapy in the treatment of ambulatory bipolar spectrum disorder with moderate-to-severe hypomania or mild mania in a randomized, double-blind, placebo-controlled, parallel group, 8-week trial in 60 outpatients with bipolar disorder, types I, II, or NOS by DSM-IV-TR criteria. Patients may have concurrent depressive and anxiety symptoms and syndromes, but not psychotic features or substance dependence. The primary outcome measure will be change in hypomanic/manic symptoms from baseline to endpoint. Secondary outcome measures will include change in depressive and anxiety symptoms, change in global severity of illness, concomitant use of adjunctive rescue anxiolytic and hypnotic medications, adherence with study medication, and degree and severity of side effects experienced.

a) Methods and Procedures This is a randomized, double-blind, placebo-controlled, parallel group, 8-week study in 60 outpatients with bipolar disorder types I, II, or NOS by DSM-IV criteria (13), whose overall bipolar illness is mild to moderately severe defined as a score of > 2 but < 5 on the CGI modified for bipolar illness [CGI-BP] (14), and who also have moderate-to-severe hypomania or mild mania, defined as a YMRS > 10 and < 21 at study entry. Subjects may have concurrent depressive or anxiety symptoms or syndromes, but they may not have psychotic features. The primary outcome measure will be change in manic symptoms as measured by the change in the Young Mania Rating Scale (YMRS)(17). Secondary outcome measures will include the Inventory for Depressive Symptoms (IDS)(18), the Hamilton Rating Scale for Anxiety (HAM-A)(20), the Clinical Global Improvement Scale modified for Bipolar Disorder (CGI-BP), the (16) Global Assessment of Functioning Scale (GAF), and the Sheehan Disability Scale (DSD)(18).

Medication Dosing:

Divalproex ER will be administered at an initial dose of 15mg/kg/day and will be titrated upward to a dose considered optimal by the investigator based on the subject's clinical response and adverse events, but not to exceed 30mg/kg/day. As needed (prn) use of lorazepam (0.5-2.0mg/day) will be allowed for the management of affective symptoms for the first two weeks of the study; prn lorazpam (0.5-1.0mg/day) will be allowed for the next 2 weeks; subsequently (for the final 4 weeks of the study), no lorazepam will be permitted. Zaleplon (10-20mg/day) will be allowed for management of insomnia throughout the study.

Screening Visit(s):

The Screening Period will last a minimum of 3 to a maximum of 30 days. At the first screening visit (Visit 0), informed consent will be obtained. The Structured Clinical Interview for DSM-IV (SCID) will be performed to establish whether the patient meets DSM-IV criteria for bipolar disorder I, II, or NOS. The YMRS(17), IDS (18), and CGI-BP (16) will be performed to establish the presence and severity of bipolar affective symptoms. If subjects are currently on psychotropic medications, these will be tapered. Subjects will need to be off any psychotropic medications for at least 1 week prior to randomization, 2 weeks if you have been taking fluoxetine and 4 weeks if you have been receiving depot antipsychotic medication. Mood charts will be administered to subjects to help them in following their symptoms. Subjects will meet with the study staff weekly during the period after they have stopped their previous psychiatric medications and before they start study medication. Medical history will be reviewed, a physical exam performed, electrocardiogram (EKG) and laboratory studies (Complete Metabolic Profile, Liver Function Tests (LFT's), CBC with diff + platelets, and Urinalysis) will be obtained. Based on these evaluations, it will be determined whether subjects meet entry criteria; subjects meeting these criteria will continue in the screening process.

Baseline Visit (last Screening Visit):

At baseline (Visit 1), subjects whose screening evaluations continue to meet all inclusion/exclusion criteria may enter the study and be randomized. Baseline ratings will be obtained, including the YMRS, IDS, HAM-A, and the Clinical Global Impression (CGI-BP). The subject must be evaluated as having modest-to-severe hypomania or mild mania on at least 2 occasions at least 3 days apart to be entered into the randomized phase. Also, the subject's bipolar disorder must be evaluated as mildly to moderately severe on at least 2 occasions at least 3 days apart, defined as a CGI-BP of > 2 and < 5, for the patient to be entered into the randomized phase. Subjects will also be evaluated with the Inventory for Depressive Symptoms (IDS), Hamilton Scale for Anxiety (HAM-A), Global Assessment of Functioning Scale - clinician rated (GAF-C), and the Sheehan Disability Scale (SDS). Blood pressure, pulse, height, and weight will be measured. Study medication will be dispensed by the Physician Investigator in the form of 500mg capsules. The dose starting range of divalproex ER will be 15 mg/kg/day.

Treatment Period:

Study visits will occur every week for the first four weeks of treatment, and then every 2 weeks until the 8th week of treatment. It is expected that divalproex ER will be adjusted to an optimal dose during the first month of treatment. The following procedures will be completed at each visit.

1. Collect unused divalproex ER and perform study drug accountability. A subject's unused study medication can be redispensed back to the subject.
2. Perform YMRS, IDS, CGI-BP, HAM-A, GAF-C, and SDS ratings.
3. Assess and record adverse events.
4. Obtain blood pressure, pulse, and weight.
5. Record concomitant medication use (from mood chart)
6. Adjust divalproex ER dose (if necessary) and dispense study drug.
7. At study visits 1,2, and 4, laboratories will be obtained (complete metabolic profile, LFT's, CBC with differential platelets, urinalysis, and serum valproate level).

Final Evaluation (week 8):

The following evaluations will be conducted at the completion of, or early withdrawal from, the 8-week treatment phase. All psychiatric evaluations and all other final study procedures (including a repeat physical exam, EKG, and laboratory studies) will be completed prior to the discontinuation of divalproex ER.

1. Collect unused divalproex ER and perform study drug accountability.
2. Assess and record adverse events.
3. Obtain blood pressure, pulse, weight, and determine BMI.
4. Perform YMRS, IDS, CGI-BP, HAM-A, GAF-C and SDS ratings.
5. Perform physical examination.
6. Obtain laboratories (Complete Metabolic Profile, LFT's, CBC with/diff + platelets, Urinalysis, and serum Valproate level).
7. Repeat EKG.
8. Record concomitant medication use (from mood chart)
9. Adjust divalproex ER dose (if necessary) and prescribe drug (if subject has responded and chooses to continue on divalproex ER), or dispense divalproex ER taper for discontinuation (if subject has not responded or if subject chooses to discontinue divalproex ER for any reason).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Subjects must have bipolar I, II, or NOS disorder as defined by DSM-IV-TR. (Bipolar NOS will include hypomania defined as in DSM-IV-TR, as well as "brief" hypomania-hypomania occurring for a duration of > 1 day but < 4 days - and antidepressant associated hypomania and mania).
3. Subjects must have moderate-to-severe hypomania or mild mania within the past 2 weeks, defined as having a YMRS >10 and < 21 at the baseline assessment.
4. Subjects' overall bipolar symptoms must be clinically significant but not greater than severe (defined as a CGI-BP >2 and < 5).
5. Subjects must be outpatients.
6. Subjects must be on no psychotropics for 1 week (2 weeks for fluoxetine and 4 weeks for depot antipsychotics) except for prn lorazepam (.5-2mg/day) or zaleplon (5-10mg qhs).
7. Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained.
8. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, intrauterine device) for at least one month prior to study entry and throughout the study.

Exclusion Criteria:

1. Subjects who do not have bipolar disorder by above DSM-IV-TR criteria.
2. Subjects whose bipolar symptoms are more than severely ill (CGI-BP > 5, YMRS > 21, or IDS > 39).
3. Subjects who are receiving treatment with an antimanic or mood stabilizing medication (lithium, valproate, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication.
4. Subjects who require hospitalization.
5. Subjects with clinically significant suicidal ideation, homicidal ideation, or psychotic features.
6. Subjects with current DSM-IV Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders or a lifetime psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
7. Subjects with DSM-IV Axis I substance dependence within the past 3 months (except for nicotine dependence).
8. Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
9. Subjects who are allergic to or who have demonstrated hypersensitivity to any valproate or divalproex preparation.
10. Women who are pregnant or nursing.
11. Subjects who have received an experimental drug or used an experimental device within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be change in hypomanic/manic symptoms from baseline to endpoint. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Martens BE, Creech RS, Welge JA, Jefferson L, Guerdjikova AI, Keck PE Jr. Randomized, double-blind, placebo-controlled study of divalproex extended release loading monotherapy in ambulatory bipolar spectrum disorder patients with moderate-to-severe hypomania or mild mania. J Clin Psychiatry. 2010 May;71(5):557-65. doi: 10.4088/JCP.08m04854yel. Epub 2010 Feb 23. PMID 20361901